CLINICAL TRIAL: NCT03252665
Title: Efficacy of Intracoronary Infusion of Different Medicine With Targeted Perfusion Catheter on Myocardial Perfusion in Patients With STEMI Undergoing Primary PCI:an Open,Prospective,Randomized,Multicenter Trial.
Brief Title: Efficacy of Intracoronary Infusion of Different Medicine in STEMI Patients Undergoing Primary PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai 10th People's Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai 6th People's Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16CR1012A
Record Dates: First submitted 2017-08-10; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: ST Segment Elevation Myocardial Infarction
Keywords: STEMI; myocardial perfusion; TMPFC; Nicorandil; Alprostadil
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Alprostadil; Nicorandil; Nitroglycerin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- alprostadil (Experimental): alprostadil,2ug, dilivered by targeted perfusion catheter in the culprit vessel after PCI in STEMI patients
  Interventions: Drug: Alprostadil
- nicorandil (Experimental): nicorandil,2mg, dilivered by targeted perfusion catheter in the culprit vessel after PCI in STEMI patients
  Interventions: Drug: Nicorandil
- nitroglycerin (Placebo Comparator): nitroglycerin,200ug, dilivered by targeted perfusion catheter in the culprit vessel after PCI in STEMI patients
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Alprostadil — alprostadil,2ug, dilivered by targeted perfusion catheter in the culprit vessel after PCI in STEMI patients
  Arms: alprostadil
Drug: Nicorandil — Nicorandil,2mg, dilivered by targeted perfusion catheter in the culprit vessel after PCI in STEMI patients
  Arms: nicorandil
Drug: Nitroglycerin — Nitroglycerin,200ug, dilivered by targeted perfusion catheter in the culprit vessel after PCI in STEMI patients
  Arms: nitroglycerin

SUMMARY:
The study intends to evaluate the efficacy of different medicine delivering by targed perfusion catheter incoronary administration on epicardial, myocardial perfusion and clinical outcomes in STEMI patients undergoing primary PCI.

DETAILED DESCRIPTION:
The goal of STEMI therapy is to successfully restore both epicardial blood flow and myocardial perfusion. PCI has been documented as being the most effective method for restoration of epicardial blood flow. However, epicardial blood flow does not necessarily equate to myocardial perfusion; not every patient with TIMI 3 flow after successful PCI achieves effective myocardial tissue-level perfusion. Although epicardial TIMI 3 flow could be restored in >90% of STEMI patients undergoing PCI, normalization of myocardial perfusion was achieved less frequently, with detrimental impacts on survival。 Currently, there are two main methods of angiographic assessment of myocardial perfusion: TIMI myocardial perfusion grading (TMPG), described by Gibson et al. and myocardial blush grading (MBG), described by Van't Hof et al. These established myocardial perfusion parameters, TMPG and MBG, have been widely used in various important trials and are reported to be highly useful in predicting clinical outcomes. However, visual assessment of these methods is categorical, subjective, and operator dependent. TIMI Myocardial Perfusion Frame Count (TMPFC), a novel and objective method that measures the filling and clearance of contrast in the myocardium using cine-angiographic frame-counting, was developed by our center to quantify myocardial tissue- level perfusion and was proved to be a predictive value on clinical prognosis.

Currently, there are two main types of interventions to improve myocardial perfusion . One kind is the mechanical method, which included thrombus aspiration catheter and the distal protective devices. It has been confirmed that the mechanical method can effectively improve epicardial and myocardial perfusion in patient with part of large vessels and high burden thrombus. But for patients with small vessels and no obvious visual thrombus, the efficacy is not significant.

The other kind intervention is medicine which included GP IIb/IIIa receptor antagonist , adenosine , sodium nitroprusside, verapamil etc. Part of the drugs have some effect but the overall clinical efficacy is still not satisfied.

The study intends to use targeted perfusion catheter to deliver drug to the distal targeted blood vessels. TMPFC and TMPG are applied to evaluate the efficacy of treatment with Nicorandil versus Alprostadil on myocardial tissue-level perfusion in STEMI patients undergoing primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Age: over 18 or 18 years old, less than 75 years old;
* Patents with myocardial infarction who have symptom onset within 6h before randomization;
* ECG: ≥2 mm ST-segment elevation in 2 contiguous precordial leads or ≥1 mm ST-segment elevation in 2 contiguous extremity leads ;
* Signed informed consent form prior to trial participation.

Exclusion Criteria:

1. Evidence of cardiac rupture;
2. ECG: new left bundle branch block;
3. Thrombolysis contradictions:
4. Severe complication

   * Other diseases with life expectancy ≤12 months;
   * Any history of Severe renal or hepatic dysfunction(hepatic failure, cirrhosis, portal hypertension and active hepatitis); Neutropenia, thrombocytopenia ; Known acute pancreatitis;
   * Known acute pericarditis and/or subacute bacterial endocarditis;
   * Arterial aneurysm, arterial/venous malformation and aorta dissection;
5. Complex heart condition

   * Cardiogenic shock(SBP <90 mmHg after fluid infusion or SBP<100 mmHg after vasoactive drugs);
   * PCI within previous 1 month or Previous coronary-artery bypass surgery(CABG);
   * Previously known multivessel coronary artery disease not suitable for revascularization;
   * Hospitalisation for cardiac reason within past 48 hours;
6. Not suitable for clinical trial

   * Inclusion in another clinical trial;
   * Previous enrolment in this study or treatment with an investigational drug or device under another study protocol in the past 7 days;
   * Pregnancy or lactating;
   * Body weight <40kg or >125kg;
   * Known hypersensitivity to any drug that may appear in the study;
   * Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
TIMI Myocardial Perfusion Frame Count (TMPFC) | One mins after PCI
  TMPFC is a novel method to standardize and quantify myocardial perfusion by timing the filling and washout of contrast in the myocardium using cine-angiographic frame-counting. Briefly, the first frame of TMPFC was defined as the frame that clearly demonstrated the first appearance of myocardial blush beyond the IRA (F1). The last frame of TMPFC was then defined as the frame where contrast or myocardial blush disappeared (F2). TMPFC is F2-F1 frame counts at a filming rate of 15 frames/sec, or (F2-F1)×2 frame counts at the corrected filming rate of 30 frames/sec
TIMI Myocardial Perfusion Frame Count (TMPFC) | One mins after intracoronary medicine infusion post-PCI
  TMPFC is a novel method to standardize and quantify myocardial perfusion by timing the filling and washout of contrast in the myocardium using cine-angiographic frame-counting. Briefly, the first frame of TMPFC was defined as the frame that clearly demonstrated the first appearance of myocardial blush beyond the IRA (F1). The last frame of TMPFC was then defined as the frame where contrast or myocardial blush disappeared (F2). TMPFC is F2-F1 frame counts at a filming rate of 15 frames/sec, or (F2-F1)×2 frame counts at the corrected filming rate of 30 frames/sec
TIMI Myocardial Perfusion Grade (TMPG) | One mins after PCI
  TMPG is an angiographic measure of myocardial perfusion
TIMI Myocardial Perfusion Grade (TMPG) | One mins after intracoronary medicine infusion post-PCI
  TMPG is an angiographic measure of myocardial perfusion

SECONDARY OUTCOMES:
ST-segment Resolution | 90 mins after PCI
  Resolution of the initial sum of ST-segment elevation ≥ 70%
Myocardial-specific isoenzyme of creatine kinase (CK-MB) enzyme levels peri-PCI | Within 0 to 48 hours after enrollment
  Infarct size is measured by the myocardial-specific isoenzyme of creatine kinase (CK-MB) area under the curve, calculated by the linear-trapezoidal method. If the baseline or last value is missing, the corresponding value will be set to zero. For missing values of intermediate time points, linear interpolation is used.
TIMI Flow Grade (TFG) | One mins after PCI
  TIMI Flow Grade (TFG)assesses flow in the epicardial arteries
TIMI Flow Grade (TFG) | One mins after intracoronary medicine infusion post-PCI
  TIMI Flow Grade (TFG)assesses flow in the epicardial arteries
TIMI Frame Count (CTFC) | One mins after PCI
  CTFC is a continuous measurement assessing flow in the epicardial arteries.
TIMI Frame Count (CTFC) | One mins after intracoronary medicine infusion post-PCI
  CTFC is a continuous measurement assessing flow in the epicardial arteries.
Wall motion score index (WMSI) and LVEF by echocardiography | Echocardiography was performed 3-5 days after PCI
  Echocardiographic index includes WMSI and LVEF
CMR defined MVO | 3-5 days post-infarct
  MVO was defined as hypoenhanced area within infracted zone measured by CMR
Infarct Size by Cardiac Magnetic Resonance Imaging (CMR) | 3-5 days post-infarct
  Infarct size (expressed as a percentage of LV myocardial mass) between two groups 3-5 days post-infarct assessed by the extent of late gadolinium enhancement on CMR

OTHER OUTCOMES:
MACE | in-hospital (within 14 days)
  MACE includes all cause death, reinfarction, target vessel revascularization, and stroke
MACE | 30 days after randomization
  MACE includes all cause death, reinfarction, target vessel revascularization, and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Ben He, MD,PhD, Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Ren Ji Hospital Afflited to School of Medicine, Shanghai Jiao Tong University, Shanghai, China

REFERENCES:
- [Background] Ding S, Pu J, Qiao ZQ, Shan P, Song W, Du Y, Shen JY, Jin SX, Sun Y, Shen L, Lim YL, He B. TIMI myocardial perfusion frame count: a new method to assess myocardial perfusion and its predictive value for short-term prognosis. Catheter Cardiovasc Interv. 2010 Apr 1;75(5):722-32. doi: 10.1002/ccd.22298. PMID 19960517
- [Background] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168
- [Background] Gibson CM, Cannon CP, Murphy SA, Ryan KA, Mesley R, Marble SJ, McCabe CH, Van De Werf F, Braunwald E. Relationship of TIMI myocardial perfusion grade to mortality after administration of thrombolytic drugs. Circulation. 2000 Jan 18;101(2):125-30. doi: 10.1161/01.cir.101.2.125. PMID 10637197
- [Background] van 't Hof AW, Liem A, Suryapranata H, Hoorntje JC, de Boer MJ, Zijlstra F. Angiographic assessment of myocardial reperfusion in patients treated with primary angioplasty for acute myocardial infarction: myocardial blush grade. Zwolle Myocardial Infarction Study Group. Circulation. 1998 Jun 16;97(23):2302-6. doi: 10.1161/01.cir.97.23.2302. PMID 9639373
- [Background] Chinese Society of Cardiology of Chinese Medical Association; Editorial Board of Chinese Journal of Cardiology. [Guideline of non-ST segment elevation acute coronary syndrome]. Zhonghua Xin Xue Guan Bing Za Zhi. 2012 May;40(5):353-67. No abstract available. Chinese. PMID 22883082
- [Background] Kidambi A, Mather AN, Motwani M, Swoboda P, Uddin A, Greenwood JP, Plein S. The effect of microvascular obstruction and intramyocardial hemorrhage on contractile recovery in reperfused myocardial infarction: insights from cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2013 Jun 27;15(1):58. doi: 10.1186/1532-429X-15-58. PMID 23806080
- [Background] Roe MT, Ohman EM, Maas AC, Christenson RH, Mahaffey KW, Granger CB, Harrington RA, Califf RM, Krucoff MW. Shifting the open-artery hypothesis downstream: the quest for optimal reperfusion. J Am Coll Cardiol. 2001 Jan;37(1):9-18. doi: 10.1016/s0735-1097(00)01101-3. PMID 11153779
- [Background] Pu J, Shan P, Ding S, Qiao Z, Jiang L, Song W, Du Y, Shen J, Shen L, Jin S, He B. Gender differences in epicardial and tissue-level reperfusion in patients undergoing primary angioplasty for acute myocardial infarction. Atherosclerosis. 2011 Mar;215(1):203-8. doi: 10.1016/j.atherosclerosis.2010.11.019. Epub 2010 Nov 26. PMID 21176835
- [Background] Pu J, Ding S, Shan P, Qiao Z, Song W, Du Y, Shen J, Jin S, He B. Comparison of epicardial and myocardial perfusions after primary coronary angioplasty for ST-elevation myocardial infarction in patients under and over 75 years of age. Aging Clin Exp Res. 2010 Aug;22(4):295-302. doi: 10.1007/BF03337726. Epub 2009 Dec 1. PMID 20009495
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Shen LH, Wan F, Shen L, Ding S, Gong XR, Qiao ZQ, Du YP, Song W, Shen JY, Jin SX, Pu J, Yao TB, Jiang LS, Li WZ, Zhou GW, Liu SW, Han YL, He B. Pharmacoinvasive therapy for ST elevation myocardial infarction in China: a pilot study. J Thromb Thrombolysis. 2012 Jan;33(1):101-8. doi: 10.1007/s11239-011-0657-7. PMID 22094974
- [Derived] Zhang W, Dai J, Zheng X, Xu K, Yang X, Shen L, Wang X, Hao Z, Qiu X, Jiang L, Shi H, Shen L, He B. Myocardial protective effect of intracoronary administration of nicorandil and alprostadil via targeted perfusion microcatheter in patients undergoing elective percutaneous coronary intervention: A randomized controlled trial. Medicine (Baltimore). 2021 Apr 16;100(15):e25551. doi: 10.1097/MD.0000000000025551. PMID 33847683